CLINICAL TRIAL: NCT01171937
Title: Risperidone Treatment In Children With Autism Spectrum Disorder And High Levels of Repetitive Behavior
Acronym: ProjectV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James McCracken, Chair, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-06-033; P50HD055784 (NIH)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Autism
Keywords: ages 8-16; Repetitive Behaviors
MeSH Terms: conditions — Autistic Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open-Label Risperidone (Active Comparator): Risperidone oral solution (1mg/mL) qd for 8 weeks.
  Interventions: Drug: Risperidone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — children get randomized to either placebo or active risperidone
  Other Names: Risperdal
  Arms: Open-Label Risperidone
Drug: Placebo — Children get randomized to either placebo or risperidone
  Other Names: Inactive medicine
  Arms: Placebo

SUMMARY:
The proposed study attempts to deepen our understanding of repetitive behaviors in autism spectrum disorders (ASD) and its treatment by examining the changes in key neural circuits associated with risperidone treatment using functional MRI. This study is a substudy of a larger center grant (IRB#07-03-066). Other studies also under this center grant, include: IRB#03-02-085, IRB#95-01-028. All participants will have the option to enter another sub-study, should they meet criteria. The proposed study will address this aim by mounting a controlled trial of 52 children with Autism Spectrum Disorder. After screening assessment, children will enter a three-part study. Phase 1 will be an 8-week, double-blind, placebo-controlled flexible dose trial of risperidone. The extension phase is a 16-week open-label maintenance phase for responders to risperidone or placebo. Non-responders to placebo will be invited to enroll in the eight-week open-label study. 48 of the participants will also undergo fMRI at Week 8 while on blinded treatment, as an optional sub-study. The medication will be dispensed in a liquid suspension and the dose will range from 0.5 mg to 4.0mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females of any race or ethnicity between the ages of 8 and 16 years,
2. Body weight greater than 20 kg body weight
3. DSM-IV diagnosis of Autistic Disorder, PDD, NOS, or Asperger's Disorder (established by clinical assessment, corroborated by standard cutoff scores on the Autism Diagnostic Interview and Autism Diagnostic Observation Schedule), as determined by ADI-R administered by raters who are trained to research reliability, and confirmed by an experienced and reliable clinician using DSM-IV-TR criteria.
4. Anticonvulsants used for the treatment of a seizure disorder will be permitted if the dosage has been stable for 4 weeks and the patient is seizure free for at least 6 months,
5. Clinical Global Impression (CGI) Severity score of at least 4; and subjects must also have a score greater than 7 on the first 3 items of the Compulsions Subscale of the Revised PDD CY-BOCS.
6. Ambulatory status (outpatient or day-treatment) at time of randomization
7. Subject must demonstrate a mental age >18 months as determined by the Vineland Adaptive Behavior Scales.
8. Subjects must be free neuroleptics two weeks prior to baseline. Subjects who are on SSRIs or stimulants, must be on a stable dose for at least 4 weeks prior to baseline visit.
9. Subjects and their parents (guardians) must be judged reliable for medication compliance and must agree to keep appointments for study visits and tests as outlined in the protocol.

Exclusion Criteria:

1. IQ below mental age of 18 months as measured by either the age-appropriate form of the Wechsler, the Revised Leiter, or the Mullen
2. Females with a positive Beta HCG pregnancy test,
3. Evidence of a prior adequate trial with risperidone (defined as duration of four weeks or more at a dose of at least 2 mg per day)
4. Evidence of hypersensitivity to risperidone (defined as allergic response [e.g., skin rash]) or potentially serious adverse effect (e.g., significant tachycardia)
5. Past history of neuroleptic malignant syndrome.
6. DSM-IV diagnosis of substance abuse.
7. A significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, or unstable seizure disorder identified by history, physical examination or laboratory tests.
8. The use of any other psychotropic medication

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James McCracken, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States